CLINICAL TRIAL: NCT02551744
Title: Pantoprazole Versus Famotidine for the Prevention of Recurrent Peptic Ulcers in Thienopyridine Users - a Double-blind Randomized Controlled Trial
Brief Title: Proton Pump Inhibitor Versus Histamine-2 Receptor Antagonist for the Prevention of Recurrent Peptic Ulcers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kaohsiung Veterans General Hospital. (Other)
Responsible Party: Principal Investigator, Ping-I (William) Hsu, M.D., Professor, Kaohsiung Veterans General Hospital.
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: VGHKS12-CT7-08
Record Dates: First submitted 2015-09-14; First posted 2015-09-16 (Estimated); Results first posted 2019-08-08 (Actual); Last update posted 2019-08-08 (Actual); Status verified 2019-06

CONDITIONS: Peptic Ulcer
Keywords: histamine-2 receptor antagonist; proton pump inhibitor; thienopyridine; clopidogrel; prevention
MeSH Terms: conditions — Peptic Ulcer | interventions — Famotidine; Pantoprazole

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- proton pump inhibitor group (Active Comparator): Pantoprazole Tab 40mg qd for 6 monthrs.
  Interventions: Drug: proton pump inhibitor group
- histamine-2 receptor antagonist group (Experimental): famotidine Tab 40 mg qd for 6 months.
  Interventions: Drug: histamine-2 receptor antagonist group

INTERVENTIONS:
Drug: histamine-2 receptor antagonist group — famotidine tab 40 mg qd for 6 months.
  Other Names: famotidine 40 mg
  Arms: histamine-2 receptor antagonist group
Drug: proton pump inhibitor group — pantoprazole tab 40 mg qd for 6 months.
  Other Names: pantoprazole 40mg
  Arms: proton pump inhibitor group

SUMMARY:
Whether pantoprazole versus famotidine for the prevention of recurrent peptic ulcers in thienopyridine users remains unclear.

DETAILED DESCRIPTION:
The aims of the randomized double-blind comparison study are to compare the efficacy of Proton Pump Inhibitor and H2 receptor antagonist for the prevention of recurrent peptic ulcers in thienopyridine users. We plan to enroll 334 thienopyridine (clopidogrel or ticlopidine) users without baseline gastroduodenal ulcer at initial endoscopy. The patients will be randomly assigned to receive either (1) pantoprazole (40 mg qd) or (2) famotidine (40 mg qd) for 6 months.The ulcer recurrence rate between the treatment groups will be compared.

ELIGIBILITY:
Inclusion Criteria:

* Recent endoscopic examination (within 2 months) reveals normal appearance or erythematous patches only (without subepithelial hemorrhages, erosions or ulcers).
* Peptic ulcers (a mucosal break ³ 5 mm in diameter) have been documented by a previous endoscopic examination.
* Subjects have received thienopyridine therapy for at least two weeks.
* Requiring long-term anti-platelet therapy for ischemic cardiovascular diseases.

Exclusion Criteria:

* A history of gastric or duodenal surgery other than oversewing of a perforation.
* Subjects who are allergic to the study drugs.
* Requiring long-term treatment with non-steroidal anti-inflammatory drugs (NSAIDs), corticosteroids, aspirin, or anticoagulant agents.
* Pregnancy.
* Subjects who have active cancer, acute serious medical illness or terminal illness.
* Subjects who have gastroesophageal reflux disease.

Ages: 20 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 101 (Actual)
Dates: Start 2012-07; Primary Completion 2018-07 (Actual); Study Completion 2018-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ping-I Hus, Bachelor, Study Chair — Kaohsiung Veterans General Hospital.
Locations (1):
- Kaohsiung Veterans General Hospital, Kaohsiung City, Taiwan

REFERENCES:
- [Background] Savi P, Nurden P, Nurden AT, Levy-Toledano S, Herbert JM. Clopidogrel: a review of its mechanism of action. Platelets. 1998;9(3-4):251-5. doi: 10.1080/09537109876799. PMID 16793712
- [Background] Boeynaems JM, van Giezen H, Savi P, Herbert JM. P2Y receptor antagonists in thrombosis. Curr Opin Investig Drugs. 2005 Mar;6(3):275-82. PMID 15816504
- [Background] Yusuf S, Zhao F, Mehta SR, Chrolavicius S, Tognoni G, Fox KK; Clopidogrel in Unstable Angina to Prevent Recurrent Events Trial Investigators. Effects of clopidogrel in addition to aspirin in patients with acute coronary syndromes without ST-segment elevation. N Engl J Med. 2001 Aug 16;345(7):494-502. doi: 10.1056/NEJMoa010746. PMID 11519503
- [Background] Bhatt DL, Fox KA, Hacke W, Berger PB, Black HR, Boden WE, Cacoub P, Cohen EA, Creager MA, Easton JD, Flather MD, Haffner SM, Hamm CW, Hankey GJ, Johnston SC, Mak KH, Mas JL, Montalescot G, Pearson TA, Steg PG, Steinhubl SR, Weber MA, Brennan DM, Fabry-Ribaudo L, Booth J, Topol EJ; CHARISMA Investigators. Clopidogrel and aspirin versus aspirin alone for the prevention of atherothrombotic events. N Engl J Med. 2006 Apr 20;354(16):1706-17. doi: 10.1056/NEJMoa060989. Epub 2006 Mar 12. PMID 16531616
- [Background] Mehta SR, Yusuf S, Peters RJ, Bertrand ME, Lewis BS, Natarajan MK, Malmberg K, Rupprecht H, Zhao F, Chrolavicius S, Copland I, Fox KA; Clopidogrel in Unstable angina to prevent Recurrent Events trial (CURE) Investigators. Effects of pretreatment with clopidogrel and aspirin followed by long-term therapy in patients undergoing percutaneous coronary intervention: the PCI-CURE study. Lancet. 2001 Aug 18;358(9281):527-33. doi: 10.1016/s0140-6736(01)05701-4. PMID 11520521
- [Background] CAPRIE Steering Committee. A randomised, blinded, trial of clopidogrel versus aspirin in patients at risk of ischaemic events (CAPRIE). CAPRIE Steering Committee. Lancet. 1996 Nov 16;348(9038):1329-39. doi: 10.1016/s0140-6736(96)09457-3. PMID 8918275
- [Background] Fork FT, Lafolie P, Toth E, Lindgarde F. Gastroduodenal tolerance of 75 mg clopidogrel versus 325 mg aspirin in healthy volunteers. A gastroscopic study. Scand J Gastroenterol. 2000 May;35(5):464-9. doi: 10.1080/003655200750023705. PMID 10868447
- [Background] Hsu PI, Lai KH, Liu CP. Esomeprazole with clopidogrel reduces peptic ulcer recurrence, compared with clopidogrel alone, in patients with atherosclerosis. Gastroenterology. 2011 Mar;140(3):791-8. doi: 10.1053/j.gastro.2010.11.056. Epub 2010 Dec 7. PMID 21144850
- [Background] Chan FK, Ching JY, Hung LC, Wong VW, Leung VK, Kung NN, Hui AJ, Wu JC, Leung WK, Lee VW, Lee KK, Lee YT, Lau JY, To KF, Chan HL, Chung SC, Sung JJ. Clopidogrel versus aspirin and esomeprazole to prevent recurrent ulcer bleeding. N Engl J Med. 2005 Jan 20;352(3):238-44. doi: 10.1056/NEJMoa042087. PMID 15659723
- [Background] Ma L, Elliott SN, Cirino G, Buret A, Ignarro LJ, Wallace JL. Platelets modulate gastric ulcer healing: role of endostatin and vascular endothelial growth factor release. Proc Natl Acad Sci U S A. 2001 May 22;98(11):6470-5. doi: 10.1073/pnas.111150798. Epub 2001 May 15. PMID 11353854
- [Background] Laine L, Maller ES, Yu C, Quan H, Simon T. Ulcer formation with low-dose enteric-coated aspirin and the effect of COX-2 selective inhibition: a double-blind trial. Gastroenterology. 2004 Aug;127(2):395-402. doi: 10.1053/j.gastro.2004.05.001. PMID 15300570
- [Background] Ng FH, Wong SY, Lam KF, Chu WM, Chan P, Ling YH, Kng C, Yuen WC, Lau YK, Kwan A, Wong BC. Famotidine is inferior to pantoprazole in preventing recurrence of aspirin-related peptic ulcers or erosions. Gastroenterology. 2010 Jan;138(1):82-8. doi: 10.1053/j.gastro.2009.09.063. Epub 2009 Nov 11. PMID 19837071
- [Background] Lanas A, Garcia-Rodriguez LA, Arroyo MT, Bujanda L, Gomollon F, Forne M, Aleman S, Nicolas D, Feu F, Gonzalez-Perez A, Borda A, Castro M, Poveda MJ, Arenas J; Investigators of the Asociacion Espanola de Gastroenterologia (AEG). Effect of antisecretory drugs and nitrates on the risk of ulcer bleeding associated with nonsteroidal anti-inflammatory drugs, antiplatelet agents, and anticoagulants. Am J Gastroenterol. 2007 Mar;102(3):507-15. doi: 10.1111/j.1572-0241.2006.01062.x. PMID 17338735
- [Background] Ng FH, Wong SY, Chang CM, Chen WH, Kng C, Lanas AI, Wong BC. High incidence of clopidogrel-associated gastrointestinal bleeding in patients with previous peptic ulcer disease. Aliment Pharmacol Ther. 2003 Aug 15;18(4):443-9. doi: 10.1046/j.1365-2036.2003.01693.x. PMID 12940930
- [Background] Laine L, Hennekens C. Proton pump inhibitor and clopidogrel interaction: fact or fiction? Am J Gastroenterol. 2010 Jan;105(1):34-41. doi: 10.1038/ajg.2009.638. Epub 2009 Nov 10. PMID 19904241
- [Background] Sibbing D, Kastrati A. Risk of combining PPIs with thienopyridines: fact or fiction? Lancet. 2009 Sep 19;374(9694):952-954. doi: 10.1016/S0140-6736(09)61562-2. Epub 2009 Aug 31. No abstract available. PMID 19726077
- [Background] Norgard NB, Mathews KD, Wall GC. Drug-drug interaction between clopidogrel and the proton pump inhibitors. Ann Pharmacother. 2009 Jul;43(7):1266-74. doi: 10.1345/aph.1M051. Epub 2009 May 26. PMID 19470853
- [Background] Simon T, Verstuyft C, Mary-Krause M, Quteineh L, Drouet E, Meneveau N, Steg PG, Ferrieres J, Danchin N, Becquemont L; French Registry of Acute ST-Elevation and Non-ST-Elevation Myocardial Infarction (FAST-MI) Investigators. Genetic determinants of response to clopidogrel and cardiovascular events. N Engl J Med. 2009 Jan 22;360(4):363-75. doi: 10.1056/NEJMoa0808227. Epub 2008 Dec 22. PMID 19106083
- [Background] Ho PM, Maddox TM, Wang L, Fihn SD, Jesse RL, Peterson ED, Rumsfeld JS. Risk of adverse outcomes associated with concomitant use of clopidogrel and proton pump inhibitors following acute coronary syndrome. JAMA. 2009 Mar 4;301(9):937-44. doi: 10.1001/jama.2009.261. PMID 19258584
- [Background] Juurlink DN, Gomes T, Ko DT, Szmitko PE, Austin PC, Tu JV, Henry DA, Kopp A, Mamdani MM. A population-based study of the drug interaction between proton pump inhibitors and clopidogrel. CMAJ. 2009 Mar 31;180(7):713-8. doi: 10.1503/cmaj.082001. Epub 2009 Jan 28. PMID 19176635
- [Background] Bhatt DL, Cryer BL, Contant CF, Cohen M, Lanas A, Schnitzer TJ, Shook TL, Lapuerta P, Goldsmith MA, Laine L, Scirica BM, Murphy SA, Cannon CP; COGENT Investigators. Clopidogrel with or without omeprazole in coronary artery disease. N Engl J Med. 2010 Nov 11;363(20):1909-17. doi: 10.1056/NEJMoa1007964. Epub 2010 Oct 6. PMID 20925534

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Proton Pump Inhibitor Group | Histamine-2 Receptor Antagonist Group
Started | 50 | 51
Completed | 50 | 51
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Proton Pump Inhibitor Group | Histamine-2 Receptor Antagonist Group | Total
Number analyzed (Participants) | 50 | 51 | 101
Age, Continuous [Mean (Standard Deviation); unit: years] | 73.1 (11.1) | 71.8 (10.9) | 72.4 (11.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 10 | 23
  Male | 37 | 41 | 78
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 50 | 51 | 101
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Taiwan | 50 | 51 | 101
history of smoking [Number; unit: participants] | 3 | 4 | 7

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Ulcer Recurrence
Description: Follow-up endoscopy was performed at the end of the 6th month
Time Frame: six month
Population: Intention to treat
Measure: Number; unit: participants
Arm/Group | Proton Pump Inhibitor Group | Histamine-2 Receptor Antagonist Group
Number analyzed (Participants) | 50 | 51
participants | 1 | 7

ADVERSE EVENTS:
Time Frame: six month
Arm/Group | Proton Pump Inhibitor Group | Histamine-2 Receptor Antagonist Group
All-Cause Mortality (participants affected / at risk) | 0/50 | 0/51
Serious Adverse Events (participants affected / at risk) | 0/50 | 0/51
Other Adverse Events (participants affected / at risk) | 1/50 | 1/51
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Proton Pump Inhibitor Group (N=50) | Histamine-2 Receptor Antagonist Group (N=51)
Abdominal pain (General disorders) | 1 (1) | 1 (1) — abdominal pain sufficient to interfere with daily life

LIMITATIONS AND CAVEATS:
The trial was performed in a single country

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol (2018-07-31): https://cdn.clinicaltrials.gov/large-docs/44/NCT02551744/Prot_000.pdf